CLINICAL TRIAL: NCT07233330
Title: Obinutuzumab Treatment in Frequently Relapsing and Rituximab-Dependent Idiopathic Nephrotic Syndrome in Adults: a Fully Academic, Single-arm, Open, Prospective, Intervention Trial
Brief Title: Obinutuzumab in Adult Rituximab-Dependent Nephrotic Syndrome
Acronym: OASIS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OASIS; 2025-523306-33-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Nephrotic Syndrome，Idiopathic
MeSH Terms: conditions — Nephrosis, Lipoid | interventions — obinutuzumab

STUDY DESIGN:
Intervention Model Description: Any included participant will serve as his/her own control. No active comparator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Obinutuzumab (Experimental): One vial of 40 mL concentrate contains 1000 mg Obinutuzumab, corresponding to a concentration before dilution of 25 mg/mL. Concentrate for solution for infusion.
  Interventions: Drug: Obinutuzumab

INTERVENTIONS:
Drug: Obinutuzumab — After induction of remission is achieved, premedication with 1000 mg of paracetamol per os and intravenous infusion of 10 mg of Chlorphenamine and 80 mg of methylprednisolone will be performed on a case to case basis The, 1000 mg of obinutuzumab diluted in 250 mL of normal saline solution will be infused at an initial rate of 50 mg/hour. After every 30 minutes, provided no adverse reaction will occur, the infusion rate will be increased by 50 mg/hour up to a maximum rate of 400 mg/hour. Vital signs will be monitored prior to the infusion, every 15 minutes during the infusion, after infusion completion and then hourly up to infusion end. Participants will be monitored for four hours after completion of drug administration and will be discharged. Then, 1000 mg of obinutuzumab diluted in 250 mL of normal saline solution will be again infused at two and four weeks after the first infusion.
  Other Names: Gazyvaro

SUMMARY:
This is a multicenter, open-label, single-arm Phase II clinical trial designed to evaluate the safety, efficacy, and immunological effects of obinutuzumab in adult patients with multi-relapsing, rituximab-dependent steroid-sensitive NS.

Obinutuzumab is a glycoengineered, humanized type II anti-CD20 monoclonal antibody that was initially developed to overcome rituximab resistance in B-cell malignancies. Obinutuzumab induced a longer and deeper B cell depletion than rituximab being able to deplete B cells in lymphoid tissue other than peripheral blood, as shown in both animal models and patients with chronic lymphocytic leukemia or kidney transplantation. Notably, obinutuzumab was found to be more efficient than rituximab in inducing B-cell cytotoxicity in-vitro, especially on naïve (IgD+CD27-) and switched (IgD-CD27+) memory B cells. This is a clinically relevant finding, because memory B cells are known to be associated with the risk of relapse after rituximab treatment in children with nephrotic syndrome. A recent retrospective study in 41 children [median (IQR) age: 10.6 (8.5-14.29) years] with steroid-dependent or frequently relapsing nephrotic syndrome, showed that treatment with obinutuzumab achieved B-cell depletion and sustained remission in 38 (93%) and 28 (68%) children at 12 and 24 months after treatment, respectively. Treatment was safe and well tolerated. Moreover, preliminary data indicate that obinutuzumab treatment can achieve complete or partial remission of the nephrotic syndrome in the large majority of adult participants with membranous nephropathy refractory to different immunosuppressive medications including rituximab, and even the human type 1 anti-CD20 antibody ofatumumab or the anti-CD38 antibody felzartamab (NCT05050214). Notably, obinutuzumab treatment achieved B-cell depletion and proteinuria reduction in all treated participants and persistent circulating anti-PLA2R antibody depletion in all participants with PLA2R-related disease even during the recovery of circulating B cells (NCT05050214). Conceivably, obinutuzumab could achieve remission of idiopathic nephrotic syndrome by inducing profound and sustained B-cell depletion, thereby inhibiting the production of anti-podocyte autoantibodies or the production of still unknown B-cell derived nephritogenic mediators and autoantibodies.

Thus, whether obinutuzumab treatment may achieve persistent remission also in adult participants with multi-relapsing, rituximab-dependent nephrotic syndrome, as previously reported in children, and as already observed in adult participants with refractory membranous nephropathy (NCT05050214), and whether this effect is associated with delayed recovery of switched memory B cells and emergence of B cells with a naïve phenotype as well as sustained reduction or depletion of circulating anti-podocyte antibodies is worth investigating.

In parallel to the evaluation of the phenotype of repopulating B cells, we will evaluate serum levels of the B-cell activating factor (BAFF). BAFF is a cytokine that orchestrates peripheral tolerance of B cells and promotes the survival of autoreactive B cells escaping central tolerance mechanisms. In participants with autoimmune diseases, such as systemic lupus erythematosus or rheumatoid arthritis, the relapse of disease activity after rituximab treatment has been associated with compensatory elevation of the B cell-activating factor BAFF levels. Elevated BAFF levels at baseline or during the follow-up may explain the resistance or dependency to anti-CD20 depleting antibodies in participants with idiopathic nephrotic syndrome.

DETAILED DESCRIPTION:
About 50% of children with steroid-sensitive nephrotic syndrome become steroid-dependent or frequently relapse. These patients may require prolonged exposure to steroids and immunosuppressive drugs over years to prevent or treat relapses, sometimes beyond adult age. The use of rituximab, a first-generation anti-CD20 monoclonal antibody, has been reported to be safe and effective in most of these cases. We found that rituximab prevented relapses of the nephrotic syndrome in approximately 50% of patients and, overall, as compared to the pre-treatment period, decreased by four-fold the incidence of relapses and reduced the need of steroid therapy to prevent and treat disease recurrences in children as well as adults with multi-relapsing, steroid-dependent idiopathic nephrotic syndrome. Finding that treatment effect was independent of the underlying pathology (minimal change disease, focal and segmental glomerulosclerosis or mesangial glomerulonephritis) suggested that in all cases the disease could be antibody-mediated and response to rituximab could be mediated by depletion of nephritogenic auto-antibodies, as previously observed in patients with PLA2R-related primary membranous nephropathy treated with rituximab. Subsequent studies found that anti-podocyte antibodiesA-B, particularly anti-nephrin antibodies, could play a key pathogenic role in the nephrotic syndrome of minimal change disease as well as of focal and segmental glomerulosclerosis. Conceivably, at least in some cases, anti-CD20 mAb therapy could achieve disease remission by inhibiting the production of these nephritogenic antibodies by autoreactive B cell clones.

Independent of the underlying pathogenetic mechanisms, most patients relapse after B-cell recovery, and some patients do not achieve B-cell depletion or relapse during peripheral B-cell depletion. Moreover, up to 30% of the patients treated with rituximab develop antidrug antibodies against rituximab, which may result in drug intolerance and/or inhibition if the patient receives further courses of rituximab.

ELIGIBILITY:
Inclusion Criteria:

* Adult age (≥18 years old)
* Rituximab-dependent idiopathic nephrotic syndrome is defined and confirmed as:

  * Availability of a recent (over the last 5 years) diagnostic kidney biopsy to confirm the diagnosis of MCD, FSGS or IgM glomerulonephritis and quantify the severity of chronic changes
  * Previous history of multi-relapsing, steroid-dependent nephrotic syndrome
  * Previous history (previous to start of the prophylactic protocol) of relapse of the nephrotic syndrome after initial complete or partial remission and further remission achieved by steroid
  * Relapse of the nephrotic syndrome within 12 months after withdrawal of rituximab prophylactic treatment defined as protein increase to >3.5g/24H P/C>3500 mg/g along with serum albumin <3.5 g/dl (A clinical, rituximab-based B-cell driven treatment protocol that, per Center practice, is aimed to prevent recurrence of the nephrotic syndrome upon re-emergence of CD20+ B cells into the circulation. Rituximab is administered as soon as B-cell counts exceed 5 cells/mm3 in at least two consecutive evaluations)
* Estimated GFR by the CKD-Epi creatinine equation (2021) ≥30 ml/min/1.73 m2
* Ability to understand and provide a valid written consent to the study according to the guidelines of the Declaration of Helsinki and Good Clinical Practice
* Compliance with an effective contraception without interruption, from 28 days before treatment start up to 18 months after treatment discontinuation, agreeing not to donate semen during treatment and for 18 months after discontinuation (if the participant is male). Furthermore, women should be advised to discontinue nursing during obinutuzumab therapy and for 18 months after the last dose of Obinutuzumab. (Please see the attached 2020 CTFG "Recommendations related to contraception and pregnancy testing in clinical trials"). Each female participant will undergo pregnancy test during the course of the study at fixed timepoints.

Exclusion Criteria:

* Concomitance of clinical conditions that could jeopardize completion of the treatment/observation period and/or confound data interpretation including:

  * Active or recent (< 5 years before enrolment) history of malignancy.
  * Other active systemic immune diseases requiring concomitant treatment with steroids or any other immunosuppressive agent
  * Severe/unstable heart failure requiring hospitalization or changes in pharmacological therapy
  * Refractory severe hypertension (BP >180/100 mmHg despite optimized pharmacological treatment with at least three blood pressure-lowering medications)
  * Recent (within the last 4 weeks) severe infections requiring hospitalization or intravenous antibiotics
  * Patients with untreated or not fully cured HCV infection
  * Planning a vaccination with live virus vaccines
  * Active bacterial, viral and/or fungal infections
  * Drug or alcohol abuse
* Pregnancy, lactation, or intention to become pregnant before or during the study period, or up to 18 months of the last dose of study treatment
* Intention to donate ova or sperm over the same time period.
* Childbearing potential without highly effective contraception methods according to the 2020 CTFG Recommendations related to contraception and pregnancy testing in clinical trials (https://www.hma.eu/fileadmin/dateien/Human_Medicines/01About_HMA/Working_Groups/CTFG/2020_09_HMA_CTFG_Contraception_guidance_Version_1.1_updated.pdf)
* Known hypersensitivity to the active ingredient or any of the excipients of the study drug
* Inability to fully understand the potential risks and benefits related to study participation
* Participation in another interventional clinical study with an investigational product since the last month before enrolment
* Any other serious medical condition, uncontrolled intercurrent illness or laboratory abnormality that, according to the investigator's judgement, would constitute an unacceptable risk of premature discontinuation from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Number of relapse-free participants | Follow-up visits, at months 2, 3, 6, 9, 12 after first drug infusion.
  Number of participants who are relapse-free for 12 months after Obinutuzumab treatment

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe L Remuzzi, M.D., Study Director — Istituto Di Ricerche Farmacologiche Mario Negri
Locations (1):
- Clinical Research Centre for Rare Diseases Aldo e Cele Daccò, Ranica, BG, Italy

IPD SHARING:
Plan to Share IPD: No